CLINICAL TRIAL: NCT01383161
Title: 18-Month Double-Blind, Placebo-Controlled Study of Curcumin
Brief Title: 18-Month Study of Memory Effects of Curcumin
Acronym: Curcumin
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Gary Small, MD, Principal Investigator, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: 11-001740; IND 112714 (Other: FDA)
Record Dates: First submitted 2011-06-22; First posted 2011-06-28 (Estimated); Results first posted 2018-03-19 (Actual); Last update posted 2020-03-03 (Actual); Status verified 2020-02

CONDITIONS: Age-associated Cognitive Impairment; Mild Cognitive Impairment (MCI)
Keywords: Curcumin; Turmeric; Memory; Cognitive Impairment; Brain Imaging; Supplement
MeSH Terms: conditions — Cognitive Dysfunction | interventions — Curcumin; Dietary Supplements; Sugars

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Curcumin (Active Comparator): Theracurmin (180mg/day)
  Interventions: Drug: Curcumin
- Placebo (Placebo Comparator): Sugar Pill
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Curcumin — Six Theracurmin capsules (containing 30 mg of curcumin each) per day for 18 months.
  Other Names: Theracurmin CR-031P™ (Dietary Supplement)
  Arms: Curcumin
Other: Placebo — Six capsules per day for 18 months.
  Other Names: Sugar Pill
  Arms: Placebo

SUMMARY:
This project is designed to study the effects of the dietary supplement curcumin on age-related cognitive impairment. In particular, the study seeks to determine the effects of curcumin on cognitive decline and the amount of abnormal amyloid protein in the brain. Genetic risk will also be studied as a potential predictor of cognitive decline.

Subjects will be randomly assigned to one of two treatment groups: either a placebo twice daily or the curcumin supplement (Theracurmin®, containing 90 mg of curcumin). The investigators expect that the volunteers receiving the curcumin supplement will show less evidence of decline after 18 months than those receiving the placebo. The investigators predict that cognitive decline and treatment response will vary according to genetic risk for Alzheimer's.

The investigators will study subjects with memory complaints aged 50-90 years. Initially, subjects will undergo a clinical assessment, an MRI and a blood draw to determine genetic risk and to rule out other neurodegenerative disorders linked to memory complaints. Subsequently, subjects will undergo an -(1-{6-[(2-[F-18]fluoroethyl)(methyl)amino]-2-naphthyl}ethylidene)malononitrile (FDDNP) PET scan and a baseline neuropsychological assessment to confirm a diagnosis of MCI or normal aging. Once enrolled, subjects will begin taking the supplement (either curcumin or a placebo). Some of the initial subjects will be asked to return every three months for regular MRIs. Every 6 months, subjects will also receive neuropsychological assessments. At the conclusion of the study, subjects will be asked to complete a final neuropsychological assessment, MRI scan, PET scan and blood draw. Additional blood will be drawn at baseline and at 18 months and frozen to assess inflammatory markers if cognitive outcomes are positive.

FDDNP-PET scans will be used to measure the amount of abnormal amyloid plaque- and tau tangle-proteins in the brain; the MRIs will be used to monitor supplement side effects and measure brain structure; the neuropsychological assessments will monitor rates of cognitive decline; the blood draws will be used to determine genetic risk and to test levels of inflammatory markers.

DETAILED DESCRIPTION:
Several lines of evidence suggest that the neuropathological and clinical decline leading to Alzheimer disease (AD) begins years before patients develop the full AD clinical syndrome (NINCDS-ADRDA diagnostic criteria; McKhann et al, 1984). Mild memory complaints build gradually years before patients develop dementia. The neuropathological hallmarks of AD, "preclinical" neuritic plaques (Braak & Braak, 1991) and neurofibrillary tangles (Price & Morris, 1999), are also present years prior to clinical diagnosis. These abnormal protein deposits correlate strongly with cognitive decline.

Preclinical amyloid deposits may begin decades prior to dementia onset. In fact, diffuse plaques in non-demented elderly persons are associated with an accelerated age-related cortical cholinergic deficit, consistent with preclinical AD (Beach et al, 1997; Arai et al, 1999). Also consistent with a prolonged preclinical disease stage is our own work showing that position emission tomography (PET) measures of cerebral glucose metabolism vary according to AD genetic risk (apolipoprotein E-4 [APOE-4]) and predict cerebral metabolic and cognitive decline in people with mild cognitive complaints (age-associated memory impairment [AAMI]; Small et al, 2000). Such observations have stimulated interest in preclinical AD markers or biomarkers of brain aging that may assist in tracking treatments of AAMI and related conditions. New PET imaging methods now make it possible to provide in vivo measures of cerebral amyloid neuritic plaques (e.g., florbetapir-PET; Clarke et al, 2011) and tau neurofibrillary tangles (e.g. FDDNP-PET; Small et al, 2006, 2009).

Despite these previous research findings, clinical trials (including those using biomarkers as response measures) and subsequent treatment recommendations have been limited to patients with the full clinical dementia syndrome or mild cognitive impairment (MCI), a condition that increases the risk for developing dementia (Petersen et al, 2001). Cholinesterase inhibitors are currently the only drugs that have FDA clearance for treatment of AD, but previous studies (e.g., Ringman et al, 2005) suggest that other interventions, such as dietary or herbal supplements, may benefit cognition, and possibly interrupt the accumulation of abnormal amyloid protein deposits in the brain. For example, curcumin (diferulomethane), a low molecular weight molecule with antioxidant and anti-inflammatory activities that is derived from dietary spice, may have both cognitive-enhancing and anti-amyloid properties (Ringman et al, 2005; Yang et al, 2005).

To address such issues, the investigators propose to build upon our group's previous longitudinal brain imaging and genetic risk studies in people with age-related memory decline. Because previous studies suggest that curcumin may improve cognitive ability and prevent the build-up of age-associated plaques and tangles in the brain, the investigators will perform a double-blind, placebo-controlled trial of curcumin to test the following hypotheses:

1. People with age-related cognitive decline (i.e., MCI, AAMI or normal aging),, who receive curcumin 90 mg twice each day will show less evidence of cognitive decline (as measured with neuropsychological assessments) than those receiving placebo after 18 months.
2. People with age-related cognitive decline who receive an oral dose of curcumin 90 mg twice each day will show less build-up of plaques and tangles (as measured with FDDNP-PET imaging) than those receiving placebo after 18 months.
3. People with age-related cognitive decline, who receive curcumin 90 mg twice each day, will show decreased measures of inflammation in the blood compared with those receiving placebo after 18 months.
4. Cognitive change, FDDNP-PET measures, and treatment response will vary according to genotypes found to influence age at dementia onset (e.g., apolipoprotein E [APOE] TOMM40).

Because curcumin may alter inflammatory markers in the blood, the investigators will draw blood samples at baseline and at 18 months and freeze them for later analyses.

To test theses hypotheses, subjects with age-related cognitive decline will be enrolled (Crook et al, 1986; Petersen et al, 2001). Subjects will be randomized, using a double-blind design, to one of two treatment groups: curcumin (three 30 mg capsules twice each day) or placebo, and followed for 18 months. FDDNP-PET scanning will be performed at baseline and at 18 months. Magnetic resonance imaging (MRI) scans also will be performed for co-registration of PET and assistance in identifying regions of interest. Neuropsychological assessments will be performed at baseline, 6 months, 12 months and at the conclusion of the clinical trial (18 months). Blood will be drawn at baseline to perform genotyping.

ELIGIBILITY:
Inclusion Criteria

1. Agreement to participate in the 18-month double-blind, placebo-controlled clinical trial of curcumin.
2. Diagnostic criteria for mild cognitive impairment (MCI) or any age related memory decline according to standard criteria (Petersen et al, 2001; Crook et al, 1986).
3. Age 50 to 90 years.
4. No significant cerebrovascular disease: modified Ischemic Score of < 4 (Rosen et al, 1980).
5. Adequate visual and auditory acuity to allow neuropsychological testing.
6. Screening laboratory tests and EKG without significant abnormalities that might interfere with the study.

Exclusion Criteria

1. Diagnosis of probable Alzheimer's disease (AD) or any other dementia (e.g., vascular, Lewy body, frontotemporal) (McKhann et al, 1984).
2. Evidence of other neurological or physical illness that can produce cognitive deterioration. Volunteers with a history of stroke, TIA, carotid bruits, or lacunes on MRI scans will be excluded.
3. Inability to undergo MRI.
4. Evidence of Parkinson's disease as determined by the motor examination (items 18-31) of the Unified Parkinson's Disease Rating Scale (Fahn et al, 1987).
5. History of myocardial infarction within the previous year, or unstable cardiac disease.
6. Uncontrolled hypertension (systolic BP > 170 or diastolic BP > 100).
7. History of significant liver disease, clinically-significant pulmonary disease, diabetes, or cancer.
8. Current diagnosis of any major psychiatric disorder according to the DSM-IV TR criteria (APA, 2000).
9. Current diagnosis or history of alcoholism or substance addiction.
10. Regular use of any medication that may affect cognitive functioning including: centrally active beta-blockers, narcotics, Clonidine, anti-Parkinsonian medications, antipsychotics, benzodiazepines, systemic corticosteroids, medications with significant cholinergic or anticholinergic effects, anti-convulsants, or Warfarin. Occasional chloral hydrate use will be allowed, but discouraged, for insomnia.
11. Use of more than one multivitamin per day. Vitamins other than the standard multivitamin supplement will not be allowed.
12. Use of medications known to affect FDDNP-PET binding (e.g., ibuprofen, naproxen).
13. Use of more than one daily baby aspirin (81mg) and/or use of any medication containing curcumin.
14. Use of cognitive enhancing supplements (e.g. Ginkgo biloba).
15. Use of any investigational drugs within the previous month or longer, depending on drug half-life.
16. Pregnancy.
17. HIV infection.
18. Evidence of vasogenic edema; specifically, evidence of more than 4 cerebral microhemorrhages (regardless of their anatomical location or diagnostic characterization as "possible" or "definite") or a single area of superficial siderosis), or evidence of a prior macrohemorrhage at screening or baseline.

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2012-03 (Actual); Primary Completion 2017-04 (Actual); Study Completion 2017-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gary W Small, MD, Principal Investigator — UCLA Longevity Center
Locations (1):
- UCLA Longevity Center, Los Angeles, California, United States

REFERENCES:
- [Background] Arai T, Ikeda K, Akiyama H, Haga C, Usami M, Sahara N, Iritani S, Mori H. A high incidence of apolipoprotein E epsilon4 allele in middle-aged non-demented subjects with cerebral amyloid beta protein deposits. Acta Neuropathol. 1999 Jan;97(1):82-4. doi: 10.1007/s004010050958. PMID 9930898
- [Background] Beach TG, Honer WG, Hughes LH. Cholinergic fibre loss associated with diffuse plaques in the non-demented elderly: the preclinical stage of Alzheimer's disease? Acta Neuropathol. 1997 Feb;93(2):146-53. doi: 10.1007/s004010050595. PMID 9039461
- [Background] Braak H, Braak E. Neuropathological stageing of Alzheimer-related changes. Acta Neuropathol. 1991;82(4):239-59. doi: 10.1007/BF00308809. PMID 1759558
- [Background] McKhann G, Drachman D, Folstein M, Katzman R, Price D, Stadlan EM. Clinical diagnosis of Alzheimer's disease: report of the NINCDS-ADRDA Work Group under the auspices of Department of Health and Human Services Task Force on Alzheimer's Disease. Neurology. 1984 Jul;34(7):939-44. doi: 10.1212/wnl.34.7.939. PMID 6610841
- [Background] Petersen RC, Stevens JC, Ganguli M, Tangalos EG, Cummings JL, DeKosky ST. Practice parameter: early detection of dementia: mild cognitive impairment (an evidence-based review) [RETIRED]. Report of the Quality Standards Subcommittee of the American Academy of Neurology. Neurology. 2001 May 8;56(9):1133-42. doi: 10.1212/wnl.56.9.1133. PMID 11342677
- [Background] Price JL, Morris JC. Tangles and plaques in nondemented aging and "preclinical" Alzheimer's disease. Ann Neurol. 1999 Mar;45(3):358-68. doi: 10.1002/1531-8249(199903)45:33.0.co;2-x. PMID 10072051
- [Background] Reiman EM, Caselli RJ, Yun LS, Chen K, Bandy D, Minoshima S, Thibodeau SN, Osborne D. Preclinical evidence of Alzheimer's disease in persons homozygous for the epsilon 4 allele for apolipoprotein E. N Engl J Med. 1996 Mar 21;334(12):752-8. doi: 10.1056/NEJM199603213341202. PMID 8592548
- [Background] Shoghi-Jadid K, Small GW, Agdeppa ED, Kepe V, Ercoli LM, Siddarth P, Read S, Satyamurthy N, Petric A, Huang SC, Barrio JR. Localization of neurofibrillary tangles and beta-amyloid plaques in the brains of living patients with Alzheimer disease. Am J Geriatr Psychiatry. 2002 Jan-Feb;10(1):24-35. PMID 11790632
- [Background] Small GW, Ercoli LM, Silverman DH, Huang SC, Komo S, Bookheimer SY, Lavretsky H, Miller K, Siddarth P, Rasgon NL, Mazziotta JC, Saxena S, Wu HM, Mega MS, Cummings JL, Saunders AM, Pericak-Vance MA, Roses AD, Barrio JR, Phelps ME. Cerebral metabolic and cognitive decline in persons at genetic risk for Alzheimer's disease. Proc Natl Acad Sci U S A. 2000 May 23;97(11):6037-42. doi: 10.1073/pnas.090106797. PMID 10811879
- [Background] Small GW, Mazziotta JC, Collins MT, Baxter LR, Phelps ME, Mandelkern MA, Kaplan A, La Rue A, Adamson CF, Chang L, et al. Apolipoprotein E type 4 allele and cerebral glucose metabolism in relatives at risk for familial Alzheimer disease. JAMA. 1995 Mar 22-29;273(12):942-7. PMID 7884953
- [Background] [No authors listed] Consensus report of the Working Group on:
- [Background] Small GW, Rabins PV, Barry PP, Buckholtz NS, DeKosky ST, Ferris SH, Finkel SI, Gwyther LP, Khachaturian ZS, Lebowitz BD, McRae TD, Morris JC, Oakley F, Schneider LS, Streim JE, Sunderland T, Teri LA, Tune LE. Diagnosis and treatment of Alzheimer disease and related disorders. Consensus statement of the American Association for Geriatric Psychiatry, the Alzheimer's Association, and the American Geriatrics Society. JAMA. 1997 Oct 22-29;278(16):1363-71. PMID 9343469
- [Background] Salloway S, Sperling R, Gilman S, Fox NC, Blennow K, Raskind M, Sabbagh M, Honig LS, Doody R, van Dyck CH, Mulnard R, Barakos J, Gregg KM, Liu E, Lieberburg I, Schenk D, Black R, Grundman M; Bapineuzumab 201 Clinical Trial Investigators. A phase 2 multiple ascending dose trial of bapineuzumab in mild to moderate Alzheimer disease. Neurology. 2009 Dec 15;73(24):2061-70. doi: 10.1212/WNL.0b013e3181c67808. Epub 2009 Nov 18. PMID 19923550
- See also: UCLA Longevity Center — http://www.semel.ucla.edu/longevity/research

RESULTS

PARTICIPANT FLOW:
Groups:
- Curcumin: Theracurmin (180mg/day)
  Curcumin: Six capsules (containing 30 mg of curcumin each) per day for 18 months.
Period: Overall Study
Arm/Group | Curcumin | Placebo
Started | 25 | 21
Completed | 20 | 17
Not Completed | 5 | 4
Not completed — Adverse Event | 5 | 1
Not completed — Withdrawal by Subject | 0 | 2
Not completed — Lack of Efficacy | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Curcumin | Placebo | Total
Number analyzed (Participants) | 25 | 21 | 46
Age, Categorical [Count of Participants; unit: Participants] — Population: Baseline numbers include all participants who completed baseline measures. Only participants for whom comparison data was obtained were included in analyses.
  Participants
    <=18 years | 0 | 0 | 0
    Between 18 and 65 years | 15 | 14 | 29
    >=65 years | 10 | 7 | 17
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.5 (8.6) | 62.5 (9.0) | 63.6 (8.8)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Baseline numbers include all participants who completed baseline measures. Only participants for whom comparison data was obtained were included in analyses.
  Participants
    Female | 16 | 11 | 27
    Male | 9 | 10 | 19
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: Baseline numbers include all participants who completed baseline measures. Only participants for whom comparison data was obtained were included in analyses.
  Participants
    Hispanic or Latino | 1 | 0 | 1
    Not Hispanic or Latino | 24 | 21 | 45
    Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: Baseline numbers include all participants who completed baseline measures. Only participants for whom comparison data was obtained were included in analyses.
  Participants
    American Indian or Alaska Native | 0 | 0 | 0
    Asian | 1 | 4 | 5
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Black or African American | 1 | 1 | 2
    White | 23 | 16 | 39
    More than one race | 0 | 0 | 0
    Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 25 | 21 | 46

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to 18 Months on Brief Visual Memory Test-Revised, Recall
Description: The Brief Visual Memory Test-Revised (BVMT-R) provides a measure of visual memory. In three learning trials, the respondent views 6 geometric figures for 10 seconds and is asked to draw as many of the figures as possible from memory in their correct location on a page in the response booklet. A Delayed Recall Trial is administered after a 25-minute delay. Recall measures standard scoring of designs for accuracy and correct placement across the three trials. Scores across the three trials are summed and range from 0 to 36, with higher scores indicating better learning. There are 6 equivalent alternate forms.
Time Frame: Baseline and 18 Months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Curcumin | Placebo
Number analyzed (Participants) | 20 | 17
units on a scale
  Baseline Cognitive Score | 19.2 (6.9) | 20.3 (6.0)
  18-Month Cognitive Score | 22.4 (6.4) | 22.5 (7.8)
Statistical Analysis 1: Comparison: Curcumin vs Placebo; Test type: Superiority; p = 0.5, mixed-effects general linear model
Statistical Analysis 2: Comparison: Curcumin; Test type: Superiority; p = 0.01, t-test, 2 sided
Statistical Analysis 3: Comparison: Placebo; Test type: Superiority; p = 0.2, t-test, 2 sided

2. Primary Outcome: Change From Baseline to 18 Months on Brief Visual Memory Test-Revised, Delay
Description: The Brief Visual Memory Test-Revised (BVMT-R) provides a measure of visual memory. In three learning trials, the respondent views 6 geometric figures for 10 seconds and is asked to draw as many of the figures as possible from memory in their correct location on a page in the response booklet. A Delayed Recall Trial is administered after a 25-minute delay. Delayed recall measures standard scoring of designs for accuracy and correct placement after delay period. Scores range from 0 to 12 and reflect recent, long-term learning, with higher scores indicating better learning. There are 6 equivalent alternate forms.
Time Frame: Baseline and 18 Months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Curcumin | Placebo
Number analyzed (Participants) | 20 | 17
units on a scale
  Baseline Cognitive Score | 7.3 (2.7) | 8.3 (2.5)
  18-Month Cognitive Score | 8.5 (2.1) | 8.5 (2.8)
Statistical Analysis 1: Comparison: Curcumin vs Placebo; Test type: Superiority; p = 0.08, mixed-effects general linear model
Statistical Analysis 2: Comparison: Curcumin; Test type: Superiority; p = .006, t-test, 2 sided
Statistical Analysis 3: Comparison: Placebo; Test type: Superiority; p = 0.8, t-test, 2 sided

3. Primary Outcome: Change From Baseline on Buschke Selective Reminding Task, Consistent Long-Term Retrieval
Description: Buschke Selective Reminding Task (SRT) is a standardized measure of verbal learning that presents 12 words to the subject who is asked to immediately recall as many words as possible. The examiner then presents words that the subject was unable to recall until the subject can recall all 12 words without prompting twice, or until the examiner has presented prompts up to 12 times. Consistent Long-Term Retrieval score is the number of words that the subject recalls without receiving prompts and indicates how well the subject consolidates the new information during the learning phase (encoding). Scores indicate the sum of consistent long-term word retrieval across the 12 trials and range from 0 to 144, with higher scores indicating better learning.
Time Frame: Baseline and 18 Months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Curcumin | Placebo
Number analyzed (Participants) | 20 | 17
units on a scale
  Baseline Cognitive Score | 72.3 (31.6) | 73.7 (31.8)
  18-Month Cognitive Score | 92.6 (30.9) | 75.6 (36.4)
Statistical Analysis 1: Comparison: Curcumin vs Placebo; Test type: Superiority; p = 0.05, mixed-effects general linear model
Statistical Analysis 2: Comparison: Curcumin; Test type: Superiority; p = 0.002, t-test, 2 sided
Statistical Analysis 3: Comparison: Placebo; Test type: Superiority; p = 0.8, t-test, 2 sided

4. Primary Outcome: Change From Baseline on Buschke Selective Reminding Task, Total Score
Description: Buschke Selective Reminding Task (SRT) is a standardized measure of verbal learning that presents 12 words to the subject who is asked to immediately recall as many words as possible. The examiner then presents words that the subject was unable to recall until the subject can recall all 12 words without prompting twice, or until the examiner has presented prompts up to 12 times. Total Recall score is the sum of words recalled over the 12 trials, which reﬂects immediate recall (short-term memory) for new information. Scores range from 0 to 144, with higher scores indicating better learning.
Time Frame: Baseline and 18 Months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Curcumin | Placebo
Number analyzed (Participants) | 20 | 17
units on a scale
  Baseline Cognitive Score | 113.7 (13.9) | 111.3 (15.6)
  18-Month Cognitive Score | 121.7 (13.2) | 112.9 (18.4)
Statistical Analysis 1: Comparison: Curcumin vs Placebo; Test type: Superiority; p = 0.08, mixed-effects general linear model
Statistical Analysis 2: Comparison: Curcumin; Test type: Superiority; p = .002, t-test, 2 sided
Statistical Analysis 3: Comparison: Placebo; Test type: Superiority; p = 0.5, t-test, 2 sided

5. Secondary Outcome: Change From Baseline to 18 Months on Trail Making Test, Part A
Description: Trail Making Test is a measure used to assess cognition and attention. Trail Making, Part A is a timed test that consists of 25 circles on a piece of paper with the numbers 1-25 written randomly in circles. The respondent is asked to draw a circle from number one, and so on, in correct numerical order, until they reach number 25. Results are reported as the number of seconds required to complete the task. Respondents were allotted as much time as necessary to complete the task. Higher scores indicate greater impairment.
Time Frame: Baseline and 18 Months
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Curcumin | Placebo
Number analyzed (Participants) | 20 | 17
seconds
  Baseline Cognitive Score | 32.6 (9.3) | 30.5 (8.3)
  18-Month Cognitive Score | 24.9 (5.3) | 28.4 (10.8)
Statistical Analysis 1: Comparison: Curcumin vs Placebo; Test type: Superiority; p = 0.04, mixed-effects general linear model
Statistical Analysis 2: Comparison: Curcumin; Test type: Superiority; p = 0.0001, t-test, 2 sided
Statistical Analysis 3: Comparison: Placebo; Test type: Superiority; p = 0.1, t-test, 2 sided

6. Secondary Outcome: Change From Baseline to 18 Months on Beck Depression Inventory (BDI)
Description: Beck Depression Inventory is a self-reported questionnaire consisting of 21 items that assess for core depressive symptoms, including sadness, sleep, suicidality, and anhedonia. Each symptom is rated from 0 (absent) to 4 (maximum severity). Total scores range from 0 (no depressive symptoms) to 84 (extreme depression), with higher scores indicating more significant depression.
Time Frame: Baseline and 18 Months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Curcumin | Placebo
Number analyzed (Participants) | 20 | 17
units on a scale
  Baseline Mood Score | 4.6 (4.5) | 4.4 (3.4)
  18-Month Mood Score | 2.7 (2.5) | 4.0 (5.0)
Statistical Analysis 1: Comparison: Curcumin vs Placebo; Test type: Superiority; p = 0.3, mixed-effects general linear model
Statistical Analysis 2: Comparison: Curcumin; Test type: Superiority; p = 0.04, t-test, 2 sided
Statistical Analysis 3: Comparison: Placebo; Test type: Superiority; p = 0.6, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: 18 months
Description: A review of possible adverse events was performed with participants every 3 months
Arm/Group | Curcumin | Placebo
All-Cause Mortality (participants affected / at risk) | 0/25 | 0/21
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/21
Other Adverse Events (participants affected / at risk) | 5/25 | 1/21
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Curcumin (N=25) | Placebo (N=21)
Gastrointestinal Complaints (Gastrointestinal disorders) | 1 (1) | 0 (0) — Participant reported single adverse event of heartburn and bloating.
Gastrointestinal Complaints (Gastrointestinal disorders) | 3 (3) | 1 (1) — General gastrointestinal complaints reported.
Abnormal MRI (Nervous system disorders) | 1 (1) | 0 (0) — Abnormal MRI unrelated to study intervention diagnosed at baseline scan.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2013-12-02): https://cdn.clinicaltrials.gov/large-docs/61/NCT01383161/Prot_SAP_000.pdf